CLINICAL TRIAL: NCT00237718
Title: Provision of Antioxidant Therapy in Hemodialysis (PATH) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050377
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Results first posted 2011-10-05 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Gamma Rays; YY1 Transcription Factor; Tocopherols; Vitamin E; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALA and Vitamin E (Active Comparator): 600 mg (2 pills 300 mg each) of alpha lipoic acid (ALA) and 666 IU (1 pill) of alpha, gamma, beta and delta (mixed) tocopherols (Vitamin E) taken orally on a daily basis for 6 months
  Interventions: Drug: Alpha, gamma, beta, and delta (mixed) tocopherols; Drug: Alpha lipoic acid
- Placebo (Placebo Comparator): placebo for ALA (2 pills) and for Vitamin E (1 pill) taken orally on a daily basis for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alpha, gamma, beta, and delta (mixed) tocopherols — approximately 666 IU daily (1 pill) for 6 months
  Other Names: Vitamin E
  Arms: ALA and Vitamin E
Drug: Alpha lipoic acid — 600 mg daily (2 pills 300 mg each) for 6 months
  Arms: ALA and Vitamin E
Drug: Placebo — placebo for alpha, gamma, beta, and delta (mixed) tocopherols; 1 pill daily for 6 months
  Arms: Placebo
Drug: Placebo — placebo for alpha lipoic acid; 2 pills daily for 6 months
  Arms: Placebo

SUMMARY:
Studies have shown that end stage renal disease (ESRD) patients have higher levels of blood markers which their body makes in response to increased stress and injury. An increase in these markers have been shown to be related to cardiovascular disease and death in ESRD patients. This study will examine whether antioxidant therapy (Vitamin E and alpha lipoic acid) may decrease these markers.

DETAILED DESCRIPTION:
Oxidative stress and acute phase inflammation are now recognized to be highly prevalent in the hemodialysis population, and several lines of evidence point to their contribution in atherosclerosis development. Biomarkers of the inflammatory state such as C-reactive protein (CRP) and interleukin-6 are robust predictors of cardiovascular events and mortality in the dialysis population. The uremic state is characterized by retention of oxidized solutes including reactive aldehyde groups and oxidized thiol groups. It has recently been demonstrated that initiation of maintenance hemodialysis does not improve biomarkers of oxidative stress or inflammation, suggesting that dialysis alone is inadequate to control the atherosclerotic uremic metabolic state. In this study we hypothesize that administration of antioxidant therapy will decrease biomarkers of acute phase inflammation and oxidative stress while improving the erythropoietic response in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end-stage renal disease receiving thrice weekly hemodialysis
2. Age > 18 years
3. Life expectancy greater than one year
4. Ability to understand and provide informed consent for participation in the study

Exclusion Criteria:

1. AIDS (HIV seropositivity is not an exclusion criteria)
2. Active malignancy excluding basal cell carcinoma of the skin
3. Gastrointestinal dysfunction requiring parenteral nutrition
4. History of functional kidney transplant < 6 months prior to study entry
5. Anticipated live donor kidney transplant over study duration
6. History of poor adherence to hemodialysis or medical regimen
7. Prisoners, patients with significant mental illness, pregnant women, and other vulnerable populations
8. Patients taking vitamin E supplements > 60 IU/day, vitamin C > 500 mg/day over the past 30 days
9. Patients taking anti-inflammatory medication except aspirin < 325 mg/day over the past 30 days
10. Patients using a temporary catheter for dialysis access
11. More than two hospitalizations within the last 90 days or one hospitalization within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — MaineHealth; Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Fresenius Medical Care North America, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Vanderbilt University Medical Center and at Fresenius Medical Care North America Dialysis clinics between April 2006 and September 2010.
Pre-assignment Details: There is a 1-month period between enrollment and assignment to a treatment group. Although 385 subjects were enrolled, only 356 were randomized (29 subjects withdrew consent prior to randomization). Also, 31 subjects were administratively withdrawn (due to widespread protocol non-compliance at one site) leaving 325 subjects assigned to a group.
Groups:
- ALA and Vitamin E: 600 mg (2 pills 300 mg each) of alpha lipoic acid (ALA) and 666 IU (1 pill) of mixed (alpha, gamma, beta and delta) tocopherols (Vitamin E) taken orally on a daily basis for 6 months
Period: Overall Study
Arm/Group | ALA and Vitamin E | Placebo
Started | 160 | 165
Completed | 114 | 124
Not Completed | 46 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALA and Vitamin E | Placebo | Total
Number analyzed (Participants) | 160 | 165 | 325
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 58 (13) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 69 | 143
  Male | 86 | 96 | 182
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 98 | 90 | 188
  White | 59 | 69 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: F2-isoprostane (F2-iso)
Description: F2-iso is a sensitive laboratory assay for serum levels of F2-isoprostane, which is a biomarker of oxidative stress.
Time Frame: month 6
Population: The number of participants for analysis was based on those subjects who completed the 6-month study. Note that 8 subjects were excluded due to samples being lost. The analysis was per protocol.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ALA and Vitamin E | Placebo
Number analyzed (Participants) | 109 | 121
ng/ml | 0.077 (0.062) | 0.073 (0.055)
Statistical Analysis 1: Comparison: ALA and Vitamin E vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

2. Secondary Outcome: Interleukin-6 (IL-6)
Description: IL-6 is a sensitive laboratory assay for serum levels of interleukin-6, which is a pro-inflammatory cytokine used to evaluate the inflammatory response.
Time Frame: month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ALA and Vitamin E | Placebo
Number analyzed (Participants) | 109 | 121
pg/ml | 19 (15) | 20 (27)
Statistical Analysis 1: Comparison: ALA and Vitamin E vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ALA and Vitamin E | Placebo
Serious Adverse Events (participants affected / at risk) | 44/160 | 52/165
Other Adverse Events (participants affected / at risk) | 91/160 | 85/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALA and Vitamin E (N=160) | Placebo (N=165)
cardiac (Cardiac disorders) | 11 (13) | 8 (13)
infection (Infections and infestations) | 7 (7) | 13 (14)
pulmonary (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (6)
GI upset (Gastrointestinal disorders) | 4 (6) | 4 (4)
access related (Vascular disorders) | 2 (4) | 4 (4) — Any adverse event related to the dialysis access (catheter, graft, or fistula).
fluid overload (Cardiac disorders) | 0 (0) | 5 (5)
diabetes (Endocrine disorders) | 1 (1) | 1 (2)
edema (Renal and urinary disorders) | 0 (0) | 1 (3)
hypertension/hypotension (Vascular disorders) | 2 (2) | 1 (1)
neurological (Nervous system disorders) | 2 (2) | 1 (1)
viral infection (Infections and infestations) | 0 (0) | 3 (3)
anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
electrolyte disorder (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
pain (General disorders) | 0 (0) | 2 (2)
dizziness (General disorders) | 0 (0) | 1 (1)
lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
trauma (General disorders) | 0 (0) | 1 (1)
other (General disorders) | 4 (4) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALA and Vitamin E (N=160) | Placebo (N=165)
GI upset (Gastrointestinal disorders) | 44 (63) | 33 (44)
infection (Infections and infestations) | 32 (38) | 36 (48)
access related (Vascular disorders) | 22 (44) | 15 (25) — Any adverse event related to the dialysis access (catheter, graft, or fistula).
pain (General disorders) | 14 (18) | 19 (27)
viral infection (Infections and infestations) | 15 (19) | 19 (22)
pulmonary (Respiratory, thoracic and mediastinal disorders) | 12 (18) | 12 (14)
cardiac (Cardiac disorders) | 12 (15) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes